CLINICAL TRIAL: NCT05989997
Title: Phase I Clinical Trial of Evaluating 68Ga-NOTA-SNA002 for the Safety Tolerance, Radiation Absorbed Dose and Dosimetry in Patients With Solid Tumor
Brief Title: Phase I Clinical Trial of 68Ga-NOTA-SNA002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SmartNuclide Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SN-SNA002-2023-001
Record Dates: First submitted 2023-07-27; First posted 2023-08-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor; Positron-Emission Tomography(PET)
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- dose escalation (Experimental): 4 subgroups mass dose escalation.
  Interventions: Drug: 68Ga-NOTA-SNA002

INTERVENTIONS:
Drug: 68Ga-NOTA-SNA002 — 68Ga-NOTA-SNA002 should be injected intravenously slowly for no less than 1min.
  Other Names: Positron Emission Tomography

SUMMARY:
The clinical trial was a single-center, dose-increasing, open trial.In this clinical trial, 68Ga-NOTA-SNA002 was injected intravenously to observe its safety tolerance, radiation absorption dose, distribution characteristics, etc. in patients with solid tumors.

DETAILED DESCRIPTION:
The study consisted of four phases: screening period , baseline period , trial period and safety follow-up period .

Screening period 2 weeks before the start of the trial, all eligible subjects were selected to participate in the clinical trial. The informed consent signed by the subjects is required before performing all the examinations in this clinical trial.

Baseline period The admission criteria were checked again, and the subjects were enrolled on the same day after the check.

Trial period Including drug administration, blood collection, image collection and pathological tissue collection.

Safe follow-up period All adverse events and drug combinations are processed and recorded during this period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including boundary values);
2. Those who have behavioral capacity, voluntarily participate in this clinical study, and sign an informed consent form (ICF);
3. Physical condition (ECOG) score 0-2 points;
4. Basal heart rate 60~100 beats/min (including the boundary value, which refers to the seated heart rate of the patient in a calm state);
5. Blood pressure measurements < High blood pressure level 1 (includes a history of high blood pressure, systolic blood pressure treated with exercise or medication; 140 and diastolic blood pressure< 90mmHg); Specialty situation
6. Patients with confirmed solid tumors (including but not limited to non-small cell lung cancer, breast cancer, head and neck squamous cell carcinoma, malignant melanoma) with or without metastatic tumors;
7. Patients whose imaging findings indicate that at least one target lesion is measurable and can be biopsied (CT, MRI, or 18F-FDG PET-CT results are acceptable);
8. Pathological findings were obtained within the previous 1 year.

Exclusion Criteria:

1. Patients who are unable to perform visits or undergo relevant examinations, operations or biopsies in accordance with the clinical trial protocol;
2. Poor nutritional status, screening BMI< 18.5, can not tolerate the test;
3. People with known or suspected evidence of active autoimmune disease (e.g., vitiligo, diabetes, residual hypothyroidism due to autoimmune disease requiring hormone replacement therapy only, autoimmunological disease such as psoriasis that does not require systemic treatment), Or diseases that are not expected to recur in the absence of external triggers are allowed to be included in the study);
4. Patients who take large doses of hormones, such as hydrocortisone or 5mg prednisone in the morning and hydrocortisone or 2.5mg prednisone in the evening;
5. Patients with serious diseases or other malignant tumors (except those who have been cured one year ago or do not require additional treatment);
6. People with known severe allergy to 68Ga-NOTA-SNA002, similar drugs or excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Safety of administration(Vital signs) | up to 7 days
  The safety of administration will be evaluated based on the assessments of blood pressure, heart rate, respiration and body temperature before and after administration(% of cases with abnormal findings relative to baseline).
Laboratory examination | up to 7 days
  such as blood routine, blood biochemistry, urine routine, coagulation function, etc., to evaluate the changes of laboratory examination of subjects before and after administration
Incidence of adverse events | through study completion, an average of 1 month
  The incident and severity of adverse events per CTCAE V5.0 criteria will be recorded following dose of 68Ga-NOTA-SNA002.
Biological distribution characteristics | 60 minutes ~120 minutes after administration
  Description of biodistribution patterns of 68Ga-NOTA-SNA002 on PET
Anti-SNA002 anti-antibody | up to 1 month
  By analyzing anti-SNA002 anti-drug antibody positive rate.

SECONDARY OUTCOMES:
Changes in whole blood and serum radioactive dose | 60 minutes after Blood sampling
  Measurement of 68Ga Radiation exposure in whole blood and serum after administration
Standardized uptake values based on whole-body PET imaging | 1 month
  Analyzing whole body PET images，Define area of interest (ROI) and/or volume of Interest (VOI), calculate standardized uptake values (SUVmax, SUVmean, etc.)
Radiation absorbed dose of major organs | 1 month
  Calculation of the radiation dose for each vital organ by means of radiation uptake values

CONTACTS AND LOCATIONS:
Overall Officials: Hongcheng Shi, Doctor, Principal Investigator — Department of Nuclear Medicine, Zhongshan Hospital, Fudan University
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No